CLINICAL TRIAL: NCT01345461
Title: Fatigability of the Quadriceps Muscle in Non-cooperating Subjects
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Jesper Poulsen, MD, Rigshospitalet, Denmark
Other Study IDs: 25428
Record Dates: First submitted 2011-04-15; First posted 2011-05-02 (Estimated); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Muscle; Fatigue; Heart
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Healthy adult volunteers: Twelve healthy adult volunteers (6 men, 6 women)
  Interventions: Device: transcutaneous electrical muscle stimulation, (model DS7A, Digitimer, Welwyn, Garden City, Hertfordshire, UK)

INTERVENTIONS:
Device: transcutaneous electrical muscle stimulation, (model DS7A, Digitimer, Welwyn, Garden City, Hertfordshire, UK) — two constant current high voltage stimulators delivered ten single stimuli twitches with biphasic square pulses at widths of 300 μs. A train generator was then switched on, triggering the delivery a 35 Hz current in bouts of 3 seconds periods separated by 1-second pause for a total of 40 tetanic contractions. In immediate succession to the tetanic contractions a second series of ten single twitch stimuli ended the protocol.
  Other Names: Health young subjects

SUMMARY:
As the critical care practice has improved over the last decades more patients are recovering from intensive care therapy. However, muscle atrophy and neuromuscular dysfunction are commonly observed sequelae after critical illness and are thought to play important roles in the development of intensive care unit acquired weakness (ICUAW). As a consequence, these entities may contribute to the impaired physical function and prolonged convalescence reported by ICU patients up to twelve months after discharge. Thus, strategies to counteract muscle atrophy and neuromuscular dysfunction acquired during the ICU stay may therefore potentially improve physical outcome and reduce the overall burden of critical illness. Limited information is available on muscle function in ICU patients and to our knowledge no muscle stimulation methods are currently available for evaluating muscle fatigue in large, proximal muscles groups, such as m. quadriceps, in non-cooperating ICU patients.

DETAILED DESCRIPTION:
Positioning of the subject: A special device, consisting of a rigid padded wooden board resting on metal bar, which was attached to the metal framing of the hospital bed, held the knee joint at a 90-degree angle and secured firm support of the entire thigh (Fig. 1). The positioning was chosen to reduce unnecessary movement and minimize risk for mechanical ventilated ICU patients. Isometric knee extension forces were therefore measured while subjects were placed in a supine position in a hospital bed with a 30-degree incline of the head and torso.

Electrical muscle stimulation: Two carbon electrode pads were placed distally over the motor point of the medial (vastus medialis) and lateral (vastus lateralis) heads of the quadriceps muscle. The motor point was defined as the location that corresponded to the lowest possible threshold current and the motor threshold current was defined as the lowest train stimulation current that resulted in visible muscle contraction. Another pair of electrodes (5x9 cm) was placed 5 cm distal to the inguinal fold (10). To optimize electrical conduction, the skin was shaved and rinsed before applying the electrodes. This approach was similar to previous studies (11).

Initially, two constant current high voltage stimulators delivered ten single stimuli twitches with biphasic square pulses at widths of 300 μs. A train generator was then switched on, triggering the delivery a 35 Hz current in bouts of 3 seconds periods separated by 1-second pause for a total of 40 tetanic contractions. In immediate succession to the tetanic contractions a second series of ten single twitch stimuli ended the protocol. Figure 2 show an example of an actual recording of the force response curve.

On the first experimental day testing current was adjusted to 75% above the motor threshold current. On the second testing day, training intensity was determined as the stimulation intensity corresponding to the same force output level (mV) as generated by the first tetanic contraction on the first testing day, while maintaining the same ratio between the medial and the lateral intensity levels.

The stimulation parameters and the two-channel stimulation method were chosen in order to increase the amount of stimulated muscle mass, ensure a safe, tetanic contraction in the non-cooperating subjects; to reduce risk of excessive muscle damage and to avoid recruitment of sensory fibers and thus minimize discomfort.

Force measurements: A height adjustable strain gauge, placed beneath the bed, were secured to the metal framing of the bed and connected horizontally (180 degree) to the subjects with a non-extensible strap placed around the angle of the subject. To minimize leg movement a second non-extensible strap were attached between the ankle and a fixed metal bar, pulling directly opposite the strap holding the strain gauge. A bridge circuit was used to detect changes in relative resistance in the strain gauge and transformed voltage changes, proportional to the torque generated by the activated muscle, were then A/D converted, sampled at 1 kHz and subsequently stored on a personal computer for further offline analysis.

Off line data analysis All motor current threshold values were the average of two measurements per side.

Tetanic contractions: To ensure attainment of plateau level of contractions torque values were calculated as the mean of the last second of the 3-s contraction. Peak tetanic torque values were the highest obtained value. The tetanic stimulation period was subdivided into five intervals where interval 1 corresponds to the first 60 seconds (1-15 contractions), interval 2 from 61-120 seconds (16-30 contractions), interval 3 from 121-160 seconds (31-40 contractions), interval 4 the first 120 seconds (1-30 contractions) and interval 5 to the total period of 160 seconds (1-40 contractions). For each interval the resistance to muscle fatigue was expressed as a Fatigue Index (FI) and calculated as the ratio between the sum of peak torque values from the final three contractions relative to the sum of peak torque values from the first three contractions. Furthermore were peak torque values for each contraction plotted and the slope of the regression line for each interval calculated.

Twitch contractions: All data were 15Hz low pass filtered and peak torque and rise-time were calculated before and after the tetanic stimulation period. For each 10-twitch series peak torque and rise-time (the slope between 30% and 70% of the twitch peak force, Nm/s) was calculated for the individual twitches. Both peak torque and rise-time were then expressed as the average values of all twitches before and after the tetanic contraction.

Data integrity:

Care was taken to ensure identical study conditions and uniformity in regard to time of day, location, equipment and procedure. Furthermore, all tests were conducted in a temperature-controlled environment with a single observer assessment and measurements regime maintained throughout the study. The same investigator (JBP), who was blinded to the intensity level, determined all threshold values and MR conducted all on-line muscle force measurements. To ensure optimal comparison between the two experimental secessions subjects were placed in a standardized position securing uniformity of posture, joint positions and orientation of the thigh. To reduce day-to-day variations in electrode placement on the thigh, these were marked, along with at least three permanent landmarks, on a transparent paper, thus serving as a "map" for a precise identification. On day seven the same investigator (JBP) then carefully replaced the electrodes identical to day 1. On both testing days, gauges were calibrated and each subject received a short standardized low intensity familiarisation session prior to the testing procedure to ensure potentiation of muscle tissue during which electrical muscle stimulation and the present protocol were carefully explained. Left/right testing order was determined after randomisation with the same order of testing maintained on the second experimental day. Subjects were instructed to be as relaxed as possible and to suppress any voluntary contraction during the test. Finally, to ensure the quality of the recorded data, knee extension forces were immediately displayed on-line on a computer screen for visual inspection.

ELIGIBILITY:
Inclusion Criteria:

healthy adult volunteers

Exclusion Criteria:

medical history of cardiovascular, metabolic or neuromuscular disorders.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: healthy adult volunteers
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Fatigue Index (ratio) | One week
  The tetanic stimulation period was subdivided into five intervals. For each interval the resistance to muscle fatigue was expressed as a Fatigue Index (FI) and calculated as the ratio between the sum of peak torque values from the final three contractions relative to the sum of peak torque values from the first three contractions.

SECONDARY OUTCOMES:
Slope of regression line (Nm/s) | One week
  Peak torque values for each contraction were plotted and the slope of the regression line for each interval calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Jesper B Poulsen, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Dept. of intensive care 4131, Rigshospitalet, Copenhagen University Hospital, Copenhagen, Denmark

REFERENCES:
- [Derived] Poulsen JB, Rose MH, Moller K, Perner A, Jensen BR. A Novel Noninvasive Method for Measuring Fatigability of the Quadriceps Muscle in Noncooperating Healthy Subjects. Biomed Res Int. 2015;2015:193493. doi: 10.1155/2015/193493. Epub 2015 Jul 21. PMID 26266252